CLINICAL TRIAL: NCT01048723
Title: A Single-arm, Open Label Phase II Study of RAD001 in Soft Tissue Extremity and/or Retroperitoneal Sarcomas
Brief Title: Study of RAD001 in Soft Tissue Extremity and/or Retroperitoneal Sarcomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis terminated funding
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15962; CRAD001CUS107T (Other: Novartis); 108182 (Other: USF IRB)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2012-07

CONDITIONS: Sarcoma
Keywords: Soft Tissue; Retroperitoneal; resectable
MeSH Terms: conditions — Sarcoma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAD001 Administration (Experimental): RAD001 was administered orally as once daily dose of 10 mg PO daily x 2 weeks (14 X 10 mg tablets) continuously from study day 1 until the end of therapy (2 weeks later) or unacceptable toxicity.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — Patients were instructed to take RAD001 in the morning, at the same time each day.
  Other Names: everolimus

SUMMARY:
The goal of this clinical research study is to learn if the study drug RAD001 can stop or slow the growth of resectable soft tissue sarcoma. The patient's physical state, their symptoms, changes in the size of the tumor, and laboratory findings obtained while on-study will help the research team decide if RAD001 is safe and effective in patients with this condition. The study drug, RAD001, is made by Novartis Pharmaceuticals Corporation.

DETAILED DESCRIPTION:
A single-arm, open label, proof of principle phase II study exploring the efficacy of RAD001 in resectable soft tissue sarcomas either in the extremities, trunk or retroperitoneum. Patients with resectable sarcomas as detailed below were to have a core biopsy for molecular markers prior to therapy with RAD001 10mg PO daily x 2 weeks. Within 7-14 days of the end of therapy with RAD001, the patients were to be brought to surgery for definitive resection or, should they be candidates for neoadjuvant radiation, would have 6 16 gauge core biopsies taken percutaneously or using image guidance. Pharmacodynamic markers as detailed in the objectives were to be assessed in the laboratory.

Patients were to be numbered sequentially from 1 to 40, or more if there were patients that dropped out due to drug toxicity, with the goal of achieving 40 patients in accrual for evaluation of the pre- and post-treatment tumor samples for Pharmacodynamic assays.

ELIGIBILITY:
Inclusion Criteria:

* Have a resectable primary or recurrent sarcoma according to diagnostic imaging criteria (computed tomography [CT] and/or magnetic resonance imaging [MRI]) that has not been previously irradiated.
* Primary/recurrent or persistent sarcoma must be amenable to core biopsy for pre RAD001 pharmacodynamic studies
* World Health Organization (WHO) performance status ≤ 2
* Adequate bone marrow function shown by: absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, Platelets ≥ 100 x 10^9/L, hemoglobin (Hb) >9 g/dL
* Adequate liver function shown by: serum bilirubin ≤ 1.5 x upper limit of normal (ULN); alanine transaminase (ALT) and aspartic transaminase (AST) ≤ 2.5x ULN
* International Normal Ratio (INR) and partial thromboplastin time (PTT) ≤1.5. (Anticoagulation allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of LMW heparin for > 2 weeks at time of randomization.)
* Adequate renal function: serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, patient can only be included after initiation of appropriate lipid lowering medication.
* Signed informed consent
* Patients with resectable soft tissue extremity or retroperitoneal sarcomas amenable to pre-treatment core biopsy
* Biopsy proven surgically resectable retroperitoneal sarcomas of any histologic grade

Exclusion Criteria:

* Currently receiving anticancer therapies or have received anticancer therapies within 4 weeks of the start of study drug. Note: Primary/recurrent/ persistent sarcoma must not have been previously treated with radiation. Primary/recurrent or persistent sarcoma must not have been treated within 4 weeks of the start of RAD001 with other chemotherapeutic agents
* Have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Should not receive immunization with attenuated live vaccines within 1 week of study entry or during study period
* Brain or leptomeningeal metastases
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: Symptomatic congestive heart failure of New York Heart Association (NYHA) Class III or IV; unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease; severely impaired lung function as defined as spirometry and diffusing lung capacity oxygenation (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air; uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN; active (acute or chronic) or uncontrolled severe infections; liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Known history of human immunodeficiency virus (HIV) seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* Patients with an active, bleeding diathesis
* Females who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of RAD001)
* Received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients
* History of noncompliance to medical regimens
* Unwilling or unable to comply with the protocol
* Cutaneous sarcomas or sarcomas where neoadjuvant chemotherapy or radiation may be indicated in the treatment plan
* Sarcomas must be deemed fully resectable by pre-treatment imaging
* No evidence of distant disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S. Zager, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 patients were to be treated with RAD001 in a neoadjuvant pre-resection manner 10mg po daily x 2 weeks with resection of their extremity or retroperitoneal tumors within 2 weeks after the conclusion of therapy. All patients with resectable sarcomas by CT or MRI imaging without evidence of distant metastases would be eligible for the trial.
Pre-assignment Details: The sarcomas must be amenable to percutaneous needle core biopsy prior to initiation of RAD001 therapy.
Period: Overall Study
Arm/Group | RAD001 Administration
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | RAD001 Administration
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Pharmacodynamics (PD) Markers
Description: PD markers of RAD001 on downstream signaling pathways in patients with sarcomas: p70S6K, S6-RP, P-AKT, cleaved PARP and PCNA by Western blot, quantitative multiplex assays and immunohistochemical studies measured pre and post the 2 week treatment of RAD001. Patients were to be separated into two groups, responders and non responders based on PD results and downstream up regulation of the referenced pathways. Mean fractional inhibition of each PD marker for the responding and non-responding groups were to be calculated. Our planned analysis was for 40 participants.
Time Frame: Pre and post the 2 week treatment
Arm/Group | RAD001 Administration
Number analyzed (Participants) | 0

2. Secondary Outcome: PD Markers (p70S6K, S6-RP, P-AKT, Cleaved PARP and PCNA)
Description: Quantitative in vivo and ex vivo assessments of PD markers (p70S6K, S6-RP, P-AKT, cleaved PARP and PCNA) were to be normalized within the same sample. The extent of inhibition is defined as the fractional inhibition in each patient calculated as [(PreRx normalized PD marker - PostRx normalized PD marker) / PreRx normalized PD marker] x 100. Same definition would apply to each of these markers. Our planned analysis was for 40 participants.
Time Frame: Post the 2 week treatment
Arm/Group | RAD001 Administration
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Pathological Response
Description: We planned to determine pathological response in terms of tumor necrosis and apoptosis assessed on the resected specimens after 2 weeks of RAD001 therapy. Percent necrosis was to be reported based on the routine H and E staining. In addition to cleaved PARP analysis, TUNEL assays were to be performed judging the amount of apoptosis in the specimens after treatment. Our planned analysis was for 40 participants.
Time Frame: Post the 2 week treatment
Arm/Group | RAD001 Administration
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Memory CD8 T Cell Enhanced Production
Description: Memory CD8 T cell enhanced production as determined by fluorescence activated cell sorter (FACS) analysis on blood and tumor core biopsy specimens taken before and after therapy with RAD001. Our planned analysis was for 40 participants.
Time Frame: Pre and Post the 2 week treatment
Arm/Group | RAD001 Administration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | RAD001 Administration
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 Administration (N=2)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis/stomatitis (Gastrointestinal disorders) | 1 (3)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated early due to sponsor budget cuts. We could not meet our accrual goal to perform planned analysis of 40 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes